CLINICAL TRIAL: NCT06374810
Title: Does Conscious Connected Breathwork Reduces Symptoms of Anxiety. A Quantitative Study Conducted in an Online Environment
Brief Title: Does Conscious Connected Breathwork Reduce Symptoms of Anxiety?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Blake (Other)
Responsible Party: Sponsor-Investigator, Richard Blake, PhD Candidate, California Institute of Integral Studies
Organization: California Institute of Integral Studies (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CCB1
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Anxiety
Keywords: anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the breathwork group or they were told that they had been placed on a waitlist and that they would participate in the 2nd cohort, which would take place after the 1st 6-week program had been completed.
  Participants in the breathwork groups were also given a 10 minute guided conscious connected breathwork recording. They were advised to do this daily to support the integration of their process. This was not mandatory. At the end of the study participants were asked how often they used the guided self-practice. The frequency of use of the self-practice was used a covariate.
Who Masked: Participant
Masking Description: Participants in group 2 were told that the trial was full but actually they were just placed in the placebo control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathwork Group (Experimental): This group participated in 6 weeks of 90-minute Conscious Connected Breathwork groups conducted via Zoom. Participants attended 1 workshop per week
  Interventions: Behavioral: Conscious Connected Breathwork
- Waitlist control group (Placebo Comparator): This group were told the 1st cohort of the study was full and they would be permitted to join cohort 2 in 6 weeks time. At the end of this waitlist period participants were invited to join the second cohort so long as they still met the inclusion criteria.
  Interventions: Other: Placebo waitlist

INTERVENTIONS:
Behavioral: Conscious Connected Breathwork — Participants were taught the Conscious Connected Breathwork Technique. 2 facilitators were monitoring and coaching the participants to ensure adherence to the technique
  Arms: Breathwork Group
Other: Placebo waitlist — Participants were told the study was full and that they were placed on a waiting list until the 1st cohort had completed the breathwork program
  Arms: Waitlist control group

SUMMARY:
The goal of this clinical trial is to test whether conscious connected breathwork reduces symptoms of anxiety in people with mild to severe anxiety symptoms, as measured by the Zung Self Rating Anxiety Scale.

The main questions aims to answer:

1. Does conscious connected breathwork reduce symptoms of anxiety?
2. Does an increased frequency of self-practice lead to even greater reductions of anxiety symptoms.

there is a comparison group: Researchers will compare whether people doing the breathwork to see if [insert effects].

Participants will participate in 1, 90 minute breath workshop per week for 6 weeks. These sessions will be held on Zoom by 2 facilitators. Participants will also be given a 10 minute recording of a guided conscious connected breathwork session that they will be encouraged to complete daily.

ELIGIBILITY:
Inclusion Criteria:

- Scores of 35 or higher on the Zung self-rating anxiety scale

Exclusion Criteria:

* anyone having completed more than 4 sessions of Conscious Connected Breathwork
* Anyone who has recently (within 1 year) started anti-depressant medication or psychotherapy
* Anyone with a history of panic disorder, psychosis, angina, pregnant, seizure disorder, glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in anxiety symptoms | 6 - 8 weeks between taking the anxiety scale either before and after the breathwork program or remaining on the wait list
  Scores on the Zung Self Rating Anxiety Scale - Scores range from a minimum of 20 and a maximum of 80. A higher score indicates more severe symptoms of anxiety than a lower score.

CONTACTS AND LOCATIONS:
Locations (1):
- CIIS, San Francisco, California, United States